CLINICAL TRIAL: NCT05371977
Title: Deep Sclerectomy Versus Trabeculectomy in Normal Tension Glaucoma
Acronym: DSTRENTG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Nina Lindbohm, Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSTRENTG
Record Dates: First submitted 2022-05-02; First posted 2022-05-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Normal Tension Glaucoma
MeSH Terms: conditions — Low Tension Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep sclerectomy (Experimental)
  Interventions: Procedure: Deep Sclerectomy
- Trabeculectomy (Active Comparator)
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Procedure: Trabeculectomy — trabeculectomy glaucoma surgery
  Arms: Trabeculectomy
Procedure: Deep Sclerectomy — deep sclerectomy glaucoma surgery
  Arms: Deep sclerectomy

SUMMARY:
The purpose of this study is to assess whether deep sclerectomy is as effective in lowering intraocular pressure (IOP) as trabeculectomy in patients with normal tension glaucoma.

DETAILED DESCRIPTION:
Subjects with normal tension glaucoma that is unstable with current medication needing filtration surgery are recruited in the study. All patients meeting the inclusion criteria and giving informed consent will be randomized to whether having deep sclerectomy or trabeculectomy.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Normal Tension Glaucoma with typical nerve fiber layer defects in red-free photographs and/or optical coherence tomography (OCT) and possible equivalent visual field defects, IOP never more than 21 mmHg, and open anterior chamber angle
* Glaucoma unstable with current medication assessed by a glaucoma specialist

Exclusion Criteria:

* Secondary Glaucoma e.g. due to previous injury or uveitis
* Exfoliation syndrome
* Pigment dispersion syndrome
* Previous transscleral or endoscopic cyclophotocoagulation
* Previous other glaucoma surgery
* Previous retinal detachment
* Previous intraocular surgery like vitrectomy and other retinal surgery
* Wet age-related macular degeneration
* Diabetic retonopathy
* Previous corneal transplant or previous refractive surgery
* Fuchs' dystrophy and other abnormalities compromising corneal clarity like scars
* The patient does not want to participate in the study
* The patient does not speak Finnish, Swedish or English
* Dementia
* Only eye with vision worse than 20/200 or loss of central visual field

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Success Rate | One year
  Decrease in Intraocular Pressure of 20 % or more or former level with fewer medications

SECONDARY OUTCOMES:
Success Rate | 5 years
  Decrease in Intraocular Pressure of 20 % or more or former level with fewer medications

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland